CLINICAL TRIAL: NCT07225920
Title: Practical Delivery of Geriatric Assessment in Community Oncology Settings (PGA)
Brief Title: Understanding Needs of Older Patients Prior to Starting Cancer Treatment
Acronym: PGA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00139618; NCI-2025-07328 (Other: NCI Trial Identifier); WF-2501CD (Other: Lead Organization Identifier); WF-2501CD (Other: DCP Identifier); WF-2501CD (Other: CTEP Identifier)
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic; Early Intervention, Educational; Educational Status; Methods; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: The primary objective of Part 1 is to refine proposed implementation strategies for delivering PGA through qualitative feedback from stakeholders. The primary objective of Part 2 is to assess the acceptability of the PGA implementation strategies, as perceived by the 3 pilot practices.
Masking Description: No Data Available
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (stakeholder interview) (Experimental): Participants from practices selected for participation in Part 1 complete a stakeholder interview (approximately 60 minutes) to gather information on current PGA relevant processes within the practice, including any anticipated barriers or facilitators to delivery, and provide feedback on proposed implementation strategies.
  Interventions: Other: Survey Administration; Other: Interview
- Part 2 (PGA education, management, and support EHR review) (Experimental): See Detailed Description
  Interventions: Other: Survey Administration; Other: Educational Intervention; Other: Assessment; Other: Internet-Based Intervention; Other: Electronic Health Record Review; Other: Interview

INTERVENTIONS:
Other: Survey Administration — Complete interest survey
Other: Interview — Complete stakeholder interview
  Arms: Part 1 (stakeholder interview)
Other: Educational Intervention — Receive provider education
  Other Names: Education for Intervention, Intervention by Education, Intervention through Education, Intervention, Educational
  Arms: Part 2 (PGA education, management, and support EHR review)
Other: Educational Intervention — Receive written and/or electronic materials on PGA delivery
  Other Names: Education for Intervention, Intervention by Education, Intervention through Education, Intervention, Educational
  Arms: Part 2 (PGA education, management, and support EHR review)
Other: Assessment — Start or increase PGA and GA management
  Other Names: Assess, Assessment, assessment, assessment, assessment, Study Assessment, Study Observation
  Arms: Part 2 (PGA education, management, and support EHR review)
Other: Internet-Based Intervention — Attend virtual meetings
  Arms: Part 2 (PGA education, management, and support EHR review)
Other: Electronic Health Record Review — Complete EHR reviews
  Arms: Part 2 (PGA education, management, and support EHR review)
Other: Survey Administration — Ancillary Studies (Patient Survey)
  Arms: Part 2 (PGA education, management, and support EHR review)
Other: Interview — Ancillary studies (Patient Interview)
  Arms: Part 2 (PGA education, management, and support EHR review)

SUMMARY:
A geriatric assessment (GA) is a structured approach to identifying and addressing the strengths and vulnerabilities of older adults with cancer. They can improve the quality of cancer care for older adults and lower side effects. It is recommended a GA be administered prior to the start of non-hormonal systemic therapy for all older adults. Despite these guidelines, only a small percentage of practices report administering them. The practical geriatric assessment (PGA) was developed to help oncology practices perform GAs. It aims to provide a brief way to evaluate older patients' physical health along with other important things like support network and impact to the patient's daily life. Typically, clinics do not receive extra training on delivering the PGA. Providing training and support for staff at cancer clinics may help deliver the enhanced PGA to older adult cancer patients who are starting a new-hormonal systemic therapy. This clinical trial looks at whether providing training and support for staff at cancer clinics can help them deliver patient check-ups (e.g., PGA) specifically designed for adults >= 65 years old (older adults) starting a new non-hormonal systemic cancer therapy. The usual approach clinics use when starting these cancer therapy courses with an older adult may vary considerably.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To refine proposed implementation strategies for delivering PGA through qualitative feedback from stakeholders. (Part 1) II. To assess the acceptability of the PGA implementation strategies, as perceived by the 3 pilot practices. (Part 2)

SECONDARY OBJECTIVES:

I. To describe current PGA relevant processes at participating practices and to describe barriers and facilitators to PGA delivery though qualitative feedback from stakeholders to help inform future implementation strategies and options for tailoring those strategies. (Part 1)

II. To assess patient participation (defined by the proportion of approached eligible patients who consent to participate and are enrolled) and patient survey response (defined by the proportion of consented patients that complete the one-time patient survey). (Part 2)

III. To assess the appropriateness of the PGA implementation strategies and the feasibility of completing the PGA with implementation strategies as perceived by the 3 pilot practices. (Part 2)

IV. To refine the process for electronic health record (EHR) data abstraction to be used in the future randomized trial. (Part 2)

V. To further evaluate the PGA process from the patient perspective to inform the future randomized trial. (Part 2)

OUTLINE: Interested Community Site practices complete the interest survey during practice recruitment and selected practices are then assigned to participate in Part 1 and/or Part 2.

PART 1: Participants from practices selected for participation in Part 1 complete a stakeholder interview (approximately 60 minutes) to gather information on current PGA relevant processes within the practice, including any anticipated barriers or facilitators to delivery, and provide feedback on proposed implementation strategies.

PART 2: Clinic Champions and available providers and staff from practices selected for participation in Part 2 will participate in a half-day orientation session with the study team, where they will receive provider education and written and/or electronic materials on PGA delivery at baseline. They will also review the current process for PGA, review the study activities and discuss strategies for implementing PGA.

Practices then start or increase PGA management to patients >= 65 years old who are starting a new non-hormonal systemic cancer therapy for 6 months. Clinic Champions also attend virtual monthly meetings (30-60 minutes) and receive active support to increase delivery of PGA for 6 months. Additionally, 15-35 patients will be provided a survey to capture their PGA experience, 4-10 patients will be asked to do an interview for further PGA details and 10-15 EHR reviews will be completed by staff per practice on these patients who received full or partial PGA on study. Finally, Clinic Champions, local providers, and staff complete a final debrief meeting to discuss the implementation of PGA in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* PART 1 ONCOLOGY CLINICIANS: Must be an oncology clinician (MDs, DOs, APPs (e.g. NP, PA)) who administers systemic therapy (chemotherapy, immunotherapy or targeted therapy).
* PART 1 ONCOLOGY CLINICIANS: Must be involved in the planning or delivery of new systemic therapies (e.g. chemotherapy, immunotherapy, targeted therapy) to patients including those >= 65 years old
* PART 1 ONCOLOGY CLINICIANS: Must be willing to participate in a semi-structured interview (approximately 60 minutes; remotely over the internet or by phone)
* PART 1 ONCOLOGY CLINICIANS: Concurrent participation in URCC-19170 is allowed, not required
* PART 1 ONCOLOGY CLINICIANS: Must be able to read, understand and speak English
* PART 1 ONCOLOGY SUPPORT STAFF STAKEHOLDER: Nurse, practice manager, or other oncology support staff who work with oncology clinicians who provide systemic therapy, help with office workflows for patient screeners, or help patients with referrals (including patients age 65 or older). May include staff that have a dual role in research and clinical support
* PART 1 ONCOLOGY SUPPORT STAFF STAKEHOLDER: Must be willing to participate in a semi-structured interview (approximately 60 minutes; remotely over the internet or by phone)
* PART 1 ONCOLOGY SUPPORT STAFF STAKEHOLDER: Concurrent participation in URCC-19170 is allowed, not required
* PART 1 ONCOLOGY SUPPORT STAFF STAKEHOLDER: Must be able to read, understand and speak English
* PART 1 PATIENT STAKEHOLDER: >= 65 years of age
* PART 1 PATIENT STAKEHOLDER: Must have initiated a new line of chemo-/immuno- and/or targeted therapy in the last 12 months
* PART 1 PATIENT STAKEHOLDER: Must be willing to participate in a semi-structured interview (approximately 60 minutes; or remotely over the internet or by phone)
* PART 1 PATIENT STAKEHOLDER: Concurrent participation in URCC-19170 is allowed, not required
* PART 1 PATIENT STAKEHOLDER: Must be able to understand and speak English
* PART 1 CAREGIVER STAKEHOLDER: Must self-report as having cared for a patient 65 years or older who initiated systemic treatment (e.g. chemo-, immuno- and/or targeted therapy) in the last 12 months. To allow for differences in how the term "caregiver" is used, we will include any family member, significant other, or friend who helps during their cancer treatment, regardless of whether they define themselves as a caregiver
* PART 1 CAREGIVER STAKEHOLDER: Must be willing to participate in a semi-structured interview (approximately 60 minutes; remotely over the internet or by phone)
* PART 1 CAREGIVER STAKEHOLDER: Concurrent participation in URCC-19170 is allowed, not required
* PART 1 CAREGIVER STAKEHOLDER: Must be able to understand and speak English
* PART 2 PRACTICE: Must be an National Cancer Institute Community Oncology Research Program (NCORP) practice (defined as one or more NCORP affiliates/sub-affiliates, which have a common administrative structure and share providers and/or patients)
* PART 2 PRACTICE: Must provide outpatient oncology care to at least 50 new patients aged 65 or over starting a new non-hormonal systemic therapy in the past 6 months
* PART 2 PRACTICE: Must have received an Introductory Email with a Practice Identification (ID) to be used to enroll the selected affiliate/sub-affiliates in Oncology Patient Enrollment Network (OPEN)
* PART 2 PRACTICE: Concurrent participation in URCC-19170 is allowed, not required
* PART 2 CLINIC CHAMPION: Must be employed in one of the selected clinics participating in the Part 2 Pilot Study
* PART 2 CLINIC CHAMPION: Must not be planning to leave their position in the next 9 months
* PART 2 CLINIC CHAMPION: Must provide care for or interact with patients age 65+ or provide administrative leadership over one of the selected clinics participating in the Part 2 Pilot Study
* PART 2 CLINIC CHAMPION: Must be willing to lead efforts to support PGA implementation within their clinic
* PART 2 CLINIC CHAMPION: Must be willing to complete the 15-minute Initial Clinic Survey at the beginning of the Part 2 Pilot Study
* PART 2 CLINIC CHAMPION: Must be willing to participate in the Initial Clinic Visit (in-person [preferred] or virtual) with the Medstar Health Research Institute (MHRI) Study Team for an estimated 60-minute in-depth discussion of the protocol. While the champion may not choose to stay with the MHRI Study Team for the rest of the half-day visit, they will facilitate plans for the other parts of the half-day site visit
* PART 2 CLINIC CHAMPION: Must be willing to participate in four 30-minute (approximately [approx.]) virtual meetings monthly during the pilot study
* PART 2 CLINIC CHAMPION: Must be willing to disseminate study materials to other relevant clinical team members, where appropriate invite the MHRI Study Team to present to other relevant clinical team members, and share updates with the MHRI Study Team during monthly virtual meetings
* PART 2 CLINIC CHAMPION: Must be willing to oversee the selection of participants to have an EHR review
* PART 2 CLINIC CHAMPION: Must be willing to participate in a 45-minute (approx.) virtual, recorded meeting at the end of the Part 2 Pilot Study (or if unavailable to attend the meeting, must be willing to complete a survey) to provide feedback on implementation strategies and on usefulness and acceptability of implementation strategies
* PART 2 CLINIC CHAMPION: Concurrent participation in URCC-19170 is allowed, not required
* PART 2 CLINIC CHAMPION: Must be able to read, understand and speak English
* PART 2 PATIENT: Must be >= 65 years of age
* PART 2 PATIENT: Must have a start date to begin a new line of cancer non-hormonal systemic therapy (i.e., chemotherapy, immunotherapy, and/or targeted therapy). The start date will be captured at OPEN enrollment
* PART 2 PATIENT: Must be willing to complete a one-time 15-minute survey
* PART 2 PATIENT: Must have completed at least one component of PGA prior to the new non-hormonal systemic therapy initiation, as identified by the local clinic provider or staff
* PART 2 PATIENT: Concurrent participation in URCC-19170 is allowed, not required
* PART 2 PATIENT: Must be able to understand and speak English
* PART 2 CLINIC DEBRIEF MEETING/SURVEY PARTICIPANTS (NOT ALREADY ENROLLED): Must work in or with the clinic that participated in Part 2 Pilot Study
* PART 2 CLINIC DEBRIEF MEETING/SURVEY PARTICIPANTS (NOT ALREADY ENROLLED): Concurrent participation in URCC-19170 is allowed, not required
* PART 2 CLINIC DEBRIEF MEETING/SURVEY PARTICIPANTS (NOT ALREADY ENROLLED): Must be able to read, understand and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative feedback on the practical geriatric assessment (PGA) implementation strategies within the context of the National Cancer Institute Community Oncology Research Program (Part 1) | Up to 6 months after the start of Part 1
  Thematic analysis will be used to identify suggested modifications that could be used to optimize acceptability of PGA implementation strategies. Intervention materials and implementation strategies will then be refined based on this feedback for further evaluation in the Part 2 Pilot Study.
Acceptability of PGA implementation strategies (Part 2) | 6 months after the start of Part 2
  Acceptability of PGA implementation strategies will be assessed qualitatively during the clinic debrief meeting for those able to attend the meeting. If a participant is unable to attend the meeting, acceptability will instead be assessed quantitatively using the Acceptability of Intervention Measure (AIM) via a REDCap survey. In this case, acceptability will be defined as a score of at least 4 on the AIM. Overall, PGA implementation strategies will be considered acceptable if the majority of participants at the debrief meeting for each clinic agree that the strategies are acceptable. If this metric is not met, strategies will be further refined before the start of the future randomized trial.

SECONDARY OUTCOMES:
Key mechanisms, intervention components, facilitators, and barriers that could inform future implementation strategies and potential modifications (Part 1) | Up to 6 months after the start of Part 1
  Thematic analysis will be used to identify key mechanisms, intervention components, facilitators, and barriers across different contextual settings that could inform future implementation strategies and potential modifications. There will be a focus on relevance for all patients and settings.
Patient participation rate (Part 2) | Up to 6 months after the start of Part 2
  A patient will be considered consented and enrolled when he or she is entered in Oncology Patient Enrollment Network. The participation rate will be calculated as the proportion of approached eligible patients (based on the WF-2501CD PGA Screening Project) who are consented and enrolled. If the participation rate is < 50%, the outreach strategies will be refined prior to starting the future randomized trial.
Patient survey response rate (Part 2) | Up to 6 months after the start of Part 2
  The one-time patient survey will be considered completed if the patient completes all survey items. The response rate will then be calculated as proportion of consented and enrolled patients who complete the survey. If the response rate is < 50%, the survey will be refined prior to starting the future randomized trial.
Appropriateness of the PGA implementation strategies (Part 2) | 6 months after the start of Part 2
  Will be assessed qualitatively during the clinic debrief meeting for those able to attend the meeting. If a participant is unable to attend the meeting, appropriateness will instead be assessed quantitatively using the Intervention Appropriateness Measure (IAM) via a REDCap survey. In this case implementation strategies will be considered appropriate if the IAM score is at least 4. If the majority of participants at the debrief meeting for each clinic do not agree on appropriateness, further refinements will be made before the start of the future randomized trial.
Feasibility of completing the PGA with implementation strategies (Part 2) | 6 months after the start of Part 2
  Will be assessed qualitatively during the clinic debrief meeting for those able to attend the meeting. If a participant is unable to attend the meeting, feasibility will instead be assessed quantitatively using the Feasibility of Intervention Measure (FIM) via a REDCap survey. In this case implementation strategies PGA will be considered feasible if the FIM score is at least 4. If the majority of participants at the debrief meeting for each clinic do not agree on feasibility, further refinements will be made before the start of the future randomized trial.
Refined electronic health record (EHR) data abstraction process (Part 2) | Up to 6 months after the start of Part 2
  To refine the process for EHR data abstraction to be used in the future randomized trial, the following data elements will be summarized: PGA domains that are documented, where in the EHR the PGA domains are documented, PGA guided actions that are documented, and where in the EHR the PGA guided actions are documented. "Raw" de-identified clinical notes will also be reviewed to confirm whether the training provided on data abstraction was sufficient.
Patient perspective of the PGA process (Part 2) | Up to 6 months after the start of Part 2
  To further evaluate the PGA process from the patient perspective to inform the future randomized trial, thematic analysis will be used to summarize the PGA experience from the patient perspective based on qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, Study Chair — Wake Forest University Health Sciences
Locations (26):
- United States (23):
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southaven, Mississippi
  - Wake Forest NCORP Research Base, Winston-Salem, North Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
- Puerto Rico (3):
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wfusm.edu
URL: http://nctn-data-archive.nci.nih.gov/